CLINICAL TRIAL: NCT07111923
Title: The Effect of Hand Position on Lower Extremity Y Balance and Reactive Balance Tests: A Cross-Sectional Study
Brief Title: The Effect of Hand Position on Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ebru Tekin, Lecturer, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023/17
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Balance Assessment; Performance
Keywords: Athlete; Balance; Hand position; Reactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance Assessment Group (Experimental)
  Interventions: Other: Balance Assesment

INTERVENTIONS:
Other: Balance Assesment — The study design was a single-group repeated measures design. Nineteen individuals meeting the inclusion criteria were included. The assessments were conducted individually in a quiet environment, isolated from other athletes and external factors. Athletes were instructed to refrain from intense exercise and training, avoid caffeine consumption, and attend the assessment in sportswear within the last 24 hours. Upon arrival for the assessments, athletes were seated to rest while demographic information was collected. Each test was explained verbally and visually, and participants were allowed to perform a trial. A crossover design method was used in the study, with the order of tests (hands on hips or hands free) determined randomly. Retest measurements were conducted 24 hours after the initial test at the same time of day. The tests performed are described below.

SUMMARY:
This study employed a single-group repeated measures design, conducted in accordance with the STROBE reporting guidelines. Nineteen participants who met the inclusion criteria were recruited. All assessments were performed individually in a quiet, controlled environment to minimize external distractions. Participants were instructed to avoid intense physical activity, caffeine consumption, and to wear appropriate sports attire for at least 48 hours prior to testing.

Upon arrival, participants rested in a seated position while demographic data were collected. Each test procedure was explained both verbally and visually, and participants were allowed to perform a practice trial to ensure comprehension. A crossover design was used to counterbalance the order of conditions (hands on hips vs. hands free), which was randomly assigned. Repeated measurements were conducted 24 hours after the initial assessments, at the same time of day, to control for diurnal variation. Detailed descriptions of the tests performed are provided in the following sections.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Female
* Volleyball player
* Age 10-18

Exclusion Criteria:

* Color blindness
* Attention deficit disorder
* Orthopedic or neurological diagnosed disease

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Y Balance Test | through study completion, an average of 1 year
  The Y Balance Test (YBT) is a shortened version of the Star Excursion Balance Test. It assesses reach distances in three directions: anterior, posteromedial, and posterolateral
Reactive Balance Test | through study completion, an average of 1 year
  The Reactive Balance Test (RBT) incorporates the YBT setup with an LED light system connected to a smartphone application. For RBT, LED lights were placed at 80% of the participants' maximum reach distance in the anterior, posteromedial, and posterolateral directions of the YBT setup (ReactionX).

SECONDARY OUTCOMES:
Lower Extremity Length | through study completion, an average of 1 year
  While the athlete was in a supine position on a mat, the distance between the ASIS (anterior superior iliac spine) and the medial malleolus was measured on both the right and left sides using a measuring tape. The lower extremity length was used to calculate the YBT composite score

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Bigadiç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No